CLINICAL TRIAL: NCT01942811
Title: US-Mexico Binational Quit Using Drugs Intervention Trial (QUIT)
Brief Title: BiNational Quit Using Drugs Intervention Trial
Acronym: BiN-QUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Lillian Gelberg, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BINAT 3P30DA027
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Drug Use; Harmful Use
Keywords: DRUG PREVENTION; BINATIONAL; CASUAL USE OF ILLICIT DRUGS; BRIEF INTERVENTION; SBIRT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The Quit Using Drugs Intervention Trial (QUIT) experimental arm includes: screening, very brief clinician advice, and telephone drug-use health education to reduce 'at risk' drug use and thus interrupt progression from casual or episodic abuse to dependence.
  Interventions: Behavioral: Quit Using Drugs Intervention Trial
- Control (No Intervention): Usual care and a health education booklet and video on cancer prevention

INTERVENTIONS:
Behavioral: Quit Using Drugs Intervention Trial — The goal of the Quit Using Drugs Intervention Trial (QUIT) is to conduct a small RCT of a primary care clinic-based very brief intervention protocol for reducing the use of illegal drugs and the occurrences of drug-related harm in low-income, racially-diverse patient populations at two 'safety-net' clinics in Los Angeles. The design will emphasize screening, very brief clinician advice, and telephone drug-use health education to reduce 'at risk' drug use and thus interrupt progression from casual or episodic abuse to dependence.
  Other Names: QUIT
  Arms: Intervention

SUMMARY:
The goal of the US-Mexico Binational Quit Using Drugs Intervention Trial (QUIT) is a multi-site study conducted in the US (East Los Angeles) and Mexico (Tijuana) which aims to reduce drug demand on both sides of the border. The study also aims to build a collaborative partnership between the US and Mexico research teams. The Bi-National QUIT Study will conduct a randomized control trial for risky drug use in several Los Angeles area community health centers. The intent of the trial is to interrupt the progression to addiction for the casual and occasional users of illicit drugs and non-medical users of pharmaceuticals. The Bi-National QUIT protocol will include (1) a computerized assessment of the patient's drug-use history (2) very brief (<5 minutes) clinician advice during a patients pre-arranged medical visit which will be preceded by a computerized assessment of the patient's drug-use history (3) a post visit assessment and video doctor (repeating the very brief clinician advice) in the waiting room (4) two post-visit telephone drug-use counseling sessions to be conducted by drug-health educators at approximately 2 and 6 weeks after the start of the intervention. Follow-up assessments will be conducted at 3 months post-randomization. Parallel activities will take place in the U.S./Los Angeles sites and Mexico/Tijuana sites. Data will be shared between both teams. Data analysis will be collaboratively conducted by both teams.

ELIGIBILITY:
Inclusion Criteria:

US Sites: Inclusion Criteria

Patients

* Adult men and women 18 and older receiving care at the study clinics
* Will be living in the LA area for the next three months
* Have a phone number at which they can be reached for the next three months
* Has a primary care visit for themselves on the date of recruitment and enrollment
* Has a primary care visit with a regular clinic provider on the date of recruitment and enrollment
* English or Spanish-speaking
* Report of drug use in the previous 90 days (i.e., cocaine or amphetamines), and has an ASSIST score between 4 and 26 indicating 'at risk' drug use
* Accessible by telephone where they can be contacted over time during the study (to conduct follow-up health education phone calls)
* Able (not cognitively impaired) and willing to cooperate with data collection and research procedures, including 2 telephone counseling sessions and 2-week, 6-week, and 3-month follow-up assessments
* Planning to be in the Los Angeles area for the next 3 months so they can complete the study period

Clinicians • Regular staff primary care clinicians of our study clinics

Mexico Sites: Inclusion Criteria

Patients

* Adult men and women 18 and older receiving care at the study clinics
* Will be living in the Tijuana area for the next three months
* Have a phone number at which they can be reached for the next three months
* Has a primary care visit for themselves on the date of recruitment and enrollment
* Has a primary care visit with a regular clinic provider on the date of recruitment and enrollment
* Spanish-speaking
* Report of drug use in the previous 90 days (i.e., cocaine or amphetamines), and has an ASSIST score between 4 and 26 indicating 'at risk' drug use
* Accessible by telephone where they can be contacted over time during the study (to conduct follow-up health education phone calls)
* Able (not cognitively impaired) and willing to cooperate with data collection and research procedures, including 2 telephone counseling sessions and 2-week, 6-week, and 3-month follow-up assessments
* Planning to be in the Tijuana area for the next 3 months so they can complete the study period

Clinicians

• Regular staff primary care clinicians of our study clinics

Exclusion Criteria:

US Sites: Exclusion Criteria

Patients

* Pregnancy. Women who report being pregnant at the time of randomization will be excluded from participation. This latter exclusion criterion is based on the following reasons: (a) The interaction of drug use (in any amount) and fetal-maternal health is physiologically complex and beyond the scope of this proposed intervention. (b) Drug users who are pregnant are considered high-risk pregnancies and will likely be lost to follow-up during the study as they will be promptly referred by their primary care clinician to an obstetrician per usual clinic protocol. However, enrolled patients who become pregnant after the intervention will not be withdrawn. Their eventual exits from the study will be counted as drop-outs and will be included as "no change" in our "intent to treat" analysis. Finally, (c) a tailored brief intervention protocol for pregnant women may require more than simple clinician advice and a 2-session phone health education program. Such an intervention would be more effective if designed around the activities of prenatal care. Previous RCTs of problem alcohol use targeting healthy adults have excluded patients who are pregnant.8,9
* Homeless status. The clinics we have chosen have large numbers of homeless patients. Since this is a study on the general poverty population, we are asking homeless status in order to avoid over-sampling homeless patients. We will set a quota on number of homeless patients we can enroll without over-sampling these patients. If we reach this quota, we will apply homeless status as an exclusion criteria for subsequent subjects.
* Repeaters. Patients who have been screened or enrolled before will be asked a set of repeater questions. This includes a question on whether they have ever been involved in our UCLA study at the clinic before. We will also ask them a set of questions that combines aspects about the potential subject (mother's first name, father's first name, month and day of birth) that will screen them out if they screen again in the future.
* ASSIST Score: Drug Dependence. The RA will receive a message that the subject scored 27+ on all illicit drugs on the WHO ASSIST (i.e. indication of possible substance dependence/addiction). The RA will inform the patient that they are at risk for certain health behaviors and ask the patient if they want to disclose this information to their doctor. If they agree to disclose information to their doctor then we will fill out a letter informing the doctor of patient's dependence on specific drugs. We will also provide the patient with a list of local substance abuse treatment referrals. Please see Appendix A for copies of these referrals (Appendix A. Los Angeles County Substance Abuse Treatment Facilities).
* From Date of Screening Subject Enrolled in a Drug Treatment Facility. Subjects enrolled in a treatment program are excluded from the study. These subjects show commitment to the treatment program. Moreover, these program would serve as a competing intervention to ours, biasing the potential effect of our intervention.

Clinicians • No exclusion criteria apply to clinicians

Mexico Sites: Exclusion Criteria

Patients

* Pregnancy. Women who report being pregnant at the time of randomization will be excluded from participation. This latter exclusion criterion is based on the following reasons: (a) The interaction of drug use (in any amount) and fetal-maternal health is physiologically complex and beyond the scope of this proposed intervention. (b) Drug users who are pregnant are considered high-risk pregnancies and will likely be lost to follow-up during the study as they will be promptly referred by their primary care clinician to an obstetrician per usual clinic protocol. However, enrolled patients who become pregnant after the intervention will not be withdrawn. Their eventual exits from the study will be counted as drop-outs and will be included as "no change" in our "intent to treat" analysis. Finally, (c) a tailored brief intervention protocol for pregnant women may require more than simple clinician advice and a 2-session phone health education program. Such an intervention would be more effective if designed around the activities of prenatal care. Previous RCTs of problem alcohol use targeting healthy adults have excluded patients who are pregnant.
* Homeless status. The clinics we have chosen have large numbers of homeless patients. Since this is a study on the general poverty population, we are asking homeless status in order to avoid over-sampling homeless patients. We will set a quota on number of homeless patients we can enroll without over-sampling these patients. If we reach this quota, we will apply homeless status as an exclusion criteria for subsequent subjects.
* Repeaters. Patients who have been screened or enrolled before will be asked a set of repeater questions. This includes a question on whether they have ever been involved in the Living Well study at the clinic before. We will also ask them a set of questions that combines aspects about the potential subject (mother's first name, father's first name, month and day of birth) that will screen them out if they screen again in the future.
* ASSIST Score: Drug Dependence. The RA will receive a message that the subject scored 27+ on all illicit drugs on the WHO ASSIST (i.e. indication of possible substance dependence/addiction). The RA will inform the patient that they are at risk for certain health behaviors and ask the patient if they want to disclose this information to their doctor. If they agree to disclose information to their doctor then we will fill out a letter informing the doctor of patient's dependence on specific drugs. We will also provide the patient with a list of local substance abuse treatment referrals.
* From Date of Screening Subject Enrolled in a Drug Treatment Facility. Subjects enrolled in a treatment program are excluded from the study. These subjects show commitment to the treatment program. Moreover, these program would serve as a competing intervention to ours, biasing the potential effect of our intervention.

Clinicians

• No exclusion criteria apply to clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Self-reported number of drug-free days at 3 months | Past 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Gelberg, MD, MSPH, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Derived] Gelberg L, Andersen RM, Rico MW, Vahidi M, Natera Rey G, Shoptaw S, Leake BD, Serota M, Singleton K, Baumeister SE. A pilot replication of QUIT, a randomized controlled trial of a brief intervention for reducing risky drug use, among Latino primary care patients. Drug Alcohol Depend. 2017 Oct 1;179:433-440. doi: 10.1016/j.drugalcdep.2017.04.022. Epub 2017 Jun 13. PMID 28844733